CLINICAL TRIAL: NCT00130754
Title: A Prospective Randomized, Controlled Pilot Study in Order to Evaluate the Place of Thymoglobuline in Non-myeloablative Allogeneic Hemapoietic Stem-cell Transplantation (NST)
Brief Title: Thymoglobuline in Non-myeloablative Allogeneic Stem-cell Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 39-14.01.05-HMO-CTIL
Record Dates: First submitted 2005-08-15; First posted 2005-08-16 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2007-11

CONDITIONS: Stem Cell Transplantation; Graft Vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Antilymphocyte Serum

ARMS (2):
- 1 (Experimental): Thymo
  Interventions: Drug: Thymoglobuline
- 2 (No Intervention)

INTERVENTIONS:
Drug: Thymoglobuline — IV 7.5 mg/kg
  Arms: 1

SUMMARY:
Allogeneic stem cell transplantation is the treatment of choice for a growing number of malignant and non-malignant indications. Until recently, myeloablative in conjunction with immunosuppressive conditioning was considered mandatory for the elimination of malignant hematopoietic cells and to prevent graft rejection. The aim of allogeneic non-myeloablative stem cell transplantation (NST) is to induce host-to-graft tolerance with fast and durable engraftment of donor stem cells, by means of conditioning, which is well-tolerated by patients. The rationale behind the NST strategy is to induce optimal graft-versus-leukemia (GVL) effects for the elimination of all malignant cells by alloreactive immunocompetent cells from a matched donor as an alternative to standard high-dose myeloablative chemo radiotherapy. The NST protocol is therefore mainly based on immunosuppression and thus contains fludarabine, low dose busulfan and anti-T-lymphocyte globulin (ATG). Thymoglobuline is a polyclonal rabbit antiserum specific for human T cells used in organ transplantation for induction of tolerance and rejection prevention and treatment. It was also used in stem-cell transplantation (SCT) for the same purposes (e.g. for generation of tolerance and rejection preclusion) as well as a treatment for graft-versus-host disease (GVHD). Data from myeloablative protocols suggest that ATG before SCT significantly reduces the risk for grade III-IV acute GVHD. This does not translate to a reduction in transplant-related mortality (TRM) because of the increased risk for infections and thus survival is unchanged. Extensive chronic GVHD was also significantly shown to be reduced in patients receiving ATG in the myeloablative setting. However, the role of ATG in the NST protocol was never evaluated in a prospective randomized trial. In view of the preliminary data suggesting of an additive effect of ATG in these circumstances we, the investigators at Hadassah Medical Organization, evaluate the effect of ATG in NST by a prospective randomized trial.

DETAILED DESCRIPTION:
Allogeneic stem cell transplantation (SCT) from a fully matched donor is the treatment of choice for a growing number of malignant and non-malignant indications. Until recently, myeloablative in conjunction with immunosuppressive conditioning was considered mandatory for the elimination of malignant hematopoietic cells and to prevent graft rejection. The aim of allogeneic non-myeloablative stem cell transplantation (NST) is to induce host-to-graft tolerance with fast and durable engraftment of donor stem cells, by means of conditioning, which is well-tolerated by patients. The rationale behind the NST strategy is to induce optimal graft-versus-leukemia (GVL) effects for the elimination of all malignant cells by alloreactive immunocompetent cells from a matched donor as an alternative to standard high-dose myeloablative chemo radiotherapy. The NST protocol is therefore mainly based on immunosuppression and thus contains fludarabine, low dose busulfan and anti-T-lymphocyte globulin (ATG). Thymoglobuline is a polyclonal rabbit antiserum specific for human T cells used in organ transplantation for induction of tolerance and rejection prevention and treatment. It was also used in SCT for the same purposes (e.g. for generation of tolerance and rejection preclusion) as well as a treatment for GVHD. Data from myeloablative protocols suggest that ATG before SCT significantly reduces the risk for grade III-IV acute GVHD. This does not translate to a reduction in TRM because of the increased risk for infections and thus survival is unchanged. Extensive chronic GVHD was also significantly shown to be reduced in patients receiving ATG in the myeloablative setting. However, the role of ATG in the NST protocol was never evaluated in a prospective randomized trial. In view of the preliminary data suggesting of an additive effect of ATG in these circumstances we propose the following clinical trial.

Objectives: To evaluate the effect of ATG vs. no ATG on the incidence of GVHD in patients undergoing NST.

Study parameters:

Primary end points -

* Acute GVHD occurrence.
* Acute GVHD grading.

Secondary end points -

* Time to acute GVHD.
* Chronic GVHD occurrence.
* Chronic GVHD grading.
* Engraftment/graft rejection
* Overall survival.
* Disease free survival.
* Infections.
* Transplant-related mortality (TRM).
* Transplant-related toxicity (TRT).

Treatment schedule:

30 patients with fully matched donors will be included. Patients will be randomized for two groups:

* Patients who will get rabbit anti-human T lymphocyte globulin (thymoglobuline R, SangStat) as a part of pre-transplant conditioning.
* Patients who will not get rabbit anti-human T lymphocyte globulin (thymoglobuline R, SangStat) as a part of pre-transplant conditioning.

Randomization:

Randomization will be done by GENZYME Israel Ltd. The center will send a randomization form to GENZYME Israel by fax and the company will fax back the randomization status of the patient. Randomization will be preformed up to day -10 pre-transplant.

Inclusion criteria:

* Patients ages 18-75 years old with a disease necessitating allogeneic SCT.
* Patients must have an HLA compatible donor willing and capable of donating peripheral blood stem cells preferably, or bone marrow progenitor cells using conventional techniques, and lymphocytes if indicated (HLA compatible defined as 5/6 or 6/6 matched related [A, B, DR] or 8/8 molecular [A, B, C, DR] matched unrelated donor).
* Both patients and donor must sign written informed consents.
* Patients must have an ECOG PS ≤ 2; Creatinine <2.0 mg/dl; Ejection fraction >40%; DLCO >50% of predicted; Serum bilirubin <3 gm/dl; elevated GPT or GOT >3 x normal values.

Exclusion criteria:

* Not fulfilling any of the inclusion criteria
* Active life-threatening infection
* Overt untreated infection
* Hypersensitivity to thymoglobuline or other rabbit produced immunoglobulin.
* HIV seropositivity, hepatitis B or C antigen positivity with active hepatitis
* Pregnant or lactating women.
* Donor contraindication (HIV seropositive confirmed by Western Blot; hepatitis B antigenemia; evidence of bone marrow disease; unable to donate bone marrow or peripheral blood due to concurrent medical condition).
* Inability to comply with study requirements.

CONDITIONING PROTOCOL:

All patients will be prepared by the NST protocol (I.V.fludarabine 30mg/m2/day [on days -10 to -5] and oral busulfan 4mg/kg in 4 divided daily doses [on days -6 and -5] or I.V. Busulfex a dose of 3.2 mg\kg on days -6 and -5,with or without I.V. ATG according to randomization group [on days -4 to -1]). ATG dosing schedule: a cumulative dose of 7.5 mg/kg ATG will be given with the following program - 0.5 mg/kg day -4, 2.0 mg/kg day -3, 2.5 mg/kg day -2, 2.5 mg/kg day -1. Each day's infusion time will be 8 hours. The last dose on day -1 should be given within 24 hours pre the stem cell infusion.

Prior to NST, all patients will receive trimethoprim/sulfamethoxazole (10 mg/kg/d trimethoprim) in days -10 to -2, acyclovir (500 mg/m2 x 3/day) from days -6 until day +100, and allopurinol (300 mg/day) on days -10 to -1. Administration of trimethoprim/sulfamethoxazole (twice weekly) will be reinstituted after recovery from neutropenia as a preventive measure against pneumocystis carinii infection. Starting on day -8, patients are monitored with a pp65 antigenemia/CMV PCR on a weekly basis to detect cytomegalovirus (CMV). Two consecutive positive PCR results or one antigenemia with more then one cell positive for pp65 serve as an indication for replacing acyclovir with ganciclovir 10 mg/kg/day until minimum of two negative tests are obtained.

Neutropenic patients with culture-negative fever receive a combination of gentamicin, cefazolin and piperacillin, as a first line antibiotic protocol. Persisting fever are treated with amikacin and tazocin as a second line protocol, while meropenem and vancomycin are used as the third line protocol. In cases of persistent fever not responding to antibiotic therapy within 5 days, amphotericin B (0.7 mg/kg/d) is added until the neutropenia resolves. No antifungal prophylaxis will be given.

Graft-vs-host disease (GVHD) prophylaxis consisting of single-drug low-dose, short- term cyclosporine- A (CSP) 3 mg/kg i.v. daily in two divided doses starting on day -4. Once the patients are mobile CSP will be administered orally. CSP dosage will be tapered during the second or third month post transplant, according to chimeric status and evidence of GVHD and then gradually stopped unless the patient will develop GVHD or graft failure. Immediately upon the appearance of signs and symptoms of GVHD, i.v. methylprednisolone (2 mg/kg) and CSP will be administered.

PBSC donors will be injected subcutaneously with granulocyte-colony stimulating factor (G-Neupogen, 5 mg/kg twice daily for 5 days) and mobilized peripheral blood stem cells will be collected on days 5 and 6.

Definitions:

Engraftment:

The 1st day of PBSC infusion is designated as "day 0". Engraftment is defined as ANC>0.5x10^9/L and peripheral WBC>1x1^09/L for 3 consecutive days and unsupported platelets>25x10^9/L.

Chimerism:

Chimerism will be assessed by standard cytogenetic analysis in male/female donor-recipient. Residual male cells in female chimera will be detected by amelogenine gene method. In sex-matched donor-recipient combinations, the various number of tandem repeats (VNTR) polymerase chain reaction (PCR) with a 5% sensitivity of detection will be used to assess the presence of residual host or donor cells.

Graft versus host disease (GVHD):

Acute and chronic GVHD will be graded according to the International Stem Cell Transplantation Registry (ISCTR) severity index.

Graft rejection:

Graft rejection is defined as peripheral blood aplasia and marrow hypoplasia > 21 days post-transplant, with no evidence of donor markers revealed by cytogenetic and molecular techniques.

Transplant-related mortality (TRM):

TRM is defined as mortality occurring due to the transplant procedure, with the patient in complete remission from the beginning of conditioning to day +100.

Transplant-related toxicity (TRT):

All nonhematological toxicities, including multi-organ dysfunction from day 0 to +100, are considered as regimen-related toxicity and graded according to the criteria of Bearman et al.

Time of follow-up: study will be ended 1-year post transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18-75 years old with a disease necessitating allogeneic SCT.
* Patients must have an HLA compatible donor willing and capable of donating peripheral blood stem cells preferably, or bone marrow progenitor cells using conventional techniques, and lymphocytes if indicated (HLA compatible defined as 5/6 or 6/6 matched related [A, B, DR] or 8/8 molecular [A, B, C, DR] matched unrelated donor).
* Both patients and donor must sign written informed consents.
* Patients must have an ECOG performance status (PS) ≤ 2; Creatinine < 2.0 mg/dl; Ejection fraction > 40%; Diffusing capacity of the lung for carbon monoxide (DLCO) > 50% of predicted; Serum bilirubin < 3 gm/dl; Elevated GPT or GOT > 3 x normal values.

Exclusion Criteria:

* Not fulfilling any of the inclusion criteria
* Active life-threatening infection
* Overt untreated infection
* Hypersensitivity to thymoglobuline or other rabbit produced immunoglobulin.
* HIV seropositivity, hepatitis B or C antigen positivity with active hepatitis
* Pregnant or lactating women.
* Donor contraindication (HIV seropositive confirmed by Western Blot; hepatitis B antigenemia; evidence of bone marrow disease; unable to donate bone marrow or peripheral blood due to concurrent medical condition).
* Inability to comply with study requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Acute GVHD occurrence | 100d
Acute GVHD grading | 100d

SECONDARY OUTCOMES:
Time to acute GVHD | 100d
Chronic GVHD occurrence | 1y
Chronic GVHD grading | 1y
Engraftment/graft rejection | 21d
Overall survival | 1y
Disease free survival | 1y
Infections | 1y
Transplant-related mortality (TRM) | 1y
Transplant-related toxicity (TRT) | 1y

CONTACTS AND LOCATIONS:
Overall Officials: Michael Y Shapira, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel